CLINICAL TRIAL: NCT07302932
Title: The Effect of Metformin Treatment on Surrogate Markers of Ageing (Leukocyte Telomere Length and Telomerase Activity), Longevity Gene Expression (Sirtuin 1, p66Shc, p53, Andmammalian Target of Rapamycin ), in North Indian Individuals With the Prediabetes: A Randomized Control Trial
Brief Title: Metformin and Molecular Aging in Prediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diabetes Foundation, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2.5/FCDOC/EC/HAO/2022-23
Record Dates: First submitted 2025-11-24; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Metformin, Prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Intervention Model Description: This clinical trial aims to evaluate the effects of metformin treatment on surrogate markers of ageing (leukocyte telomere length and telomerase activity), in the setting of pre-diabetes. We intend to compare treatment with metformin for six months, versus placebo in pre-diabetic subjects. We will assess the surrogate markers of ageing (leukocyte telomere length and telomerase activity) and the expression of longevity genes SIRT1, p66Shc, p53 and mTOR in peripheral blood mononuclear cells (PBMCs) before and after 6 months of metformin treatment.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients were recruited from Fortis C-DOC OPD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- placebo for six months (Experimental): Following a two-week diet and exercise run-in period, subjects will be randomized to receive either metformin (500mg twice daily after meals) or matching placebo for six months. All participants will monitor fasting and postprandial blood glucose (post-breakfast, post-lunch, post-dinner) monthly at home using a glucose meter. Both groups will maintain daily diaries recording tablet consumption and any missed doses. A three-month medication supply will be provided at each visit, with leftover tablets counted to assess compliance.
  Interventions: Drug: Metformin treatment
- Effect of metformin treatment on Leukocyte telomere length (Experimental): Analyzed by qPCR for T/S ratio.
  Interventions: Drug: Metformin treatment; Drug: Analyzed by qPCR for T/S ratio.
- To evaluate the effects of metformin treatment on telomerase activity (Experimental): Telomerase activity was done by ELISA Mathod
  Interventions: Drug: Metformin treatment
- Expression of longevity genes SIRT1, p66Shc, p53 and mTOR (Experimental): Investigators were assessed the expression of longevity genes SIRT1, p66Shc, p53 and mTOR in peripheral blood mononuclear cells (PBMCs) before and after 6 months of metformin treatment.
  Interventions: Drug: Metformin treatment

INTERVENTIONS:
Drug: Metformin treatment — A computer-generated randomization sequence will be created by an independent statistician using an unrestricted scheme. Allocation will be concealed in serially numbered, sealed, opaque envelopes held by non-study office staff.
  After a two-week diet and exercise run-in period, subjects will be randomized to receive either metformin (500mg twice daily) or placebo for six months. Participants will monitor fasting and postprandial blood glucose monthly at home. Medication adherence will be tracked through daily diaries and pill counts at three-month visits.
  Compliance (target ≥85%) will be maintained through biweekly phone calls (urban areas), bi-monthly home visits by health workers (rural areas), and three-monthly motivational sessions.
  Other Names: Placebo
Drug: Analyzed by qPCR for T/S ratio. — Analyzed by qPCR for T/S ratio.
  Arms: Effect of metformin treatment on Leukocyte telomere length

SUMMARY:
The incidence and prevalence of type 2 diabetes mellitus (T2DM) are increasing globally. The global prevalence of diabetes has nearly doubled since 1980, rising from 4.7% to 8.5% in the adult population. Asian Indians have one of the highest incidence rates of pre-diabetes (10.3%) and type 2 diabetes mellitus (T2DM) (8.8%) among all major ethnic groups, and the conversion from pre-diabetes to diabetes occurs more rapidly in this population.

Metformin has been shown to effectively prevent the progression of prediabetes to overt diabetes. Furthermore, metformin improves lifespan in animal models through an anti-ageing pathway driven by mTOR. Metformin has also been shown to protect endothelial cells from hyperglycaemic damage by directly stimulating the expression of Sirtuin-1 (SIRT1), a deacetylase involved in metabolism and longevity by modulating SIRT1 downstream targets FoxO1 and p53/p21. It is important to note thatSIRT1, andmammalian target of rapamycin (mTOR) form a network that connects cellular metabolism and longevity programmes.

Only one study is available which has explored the relationship of metformin with longevity. Previous study conducted a single-blind randomized placebo-controlled trial in prediabetic subjects in Italy (n, 38) who received metformin 1500mg/day (n, 19) or placebo (n, 19) for 2 months. They demonstrated that metformin use significantly increased insulin sensitivity and metabolic parameters, SIRT1 gene/protein expression, and SIRT1 promoter chromatin accessibility. They also demonstrated that metformin use increased mTOR gene expression with a concurrent decrease in p70S6K phosphorylation and altered the plasma N-glycan profile. These authors concluded that in individuals with prediabetes, metformin ameliorated effector pathways that have been shown to regulate longevity in animal models.

The investigators recently did a study on 797 prediabetic women from north India (492 of whom were obese). In this study the investigators reported that age, obesity, and subcutaneous adiposity (predominantly truncal) are the main causes of leukocyte telomere shortening. It is yet unknown how metformin impacts aging-related genes and surrogate markers of ageing in the Asian Indian population.

This clinical trial aims to evaluate the effects of metformin treatment on surrogate markers of ageing (leukocyte telomere length and telomerase activity), in the setting of pre-diabetes. We intend to compare treatment with metformin for six months, versus placebo in pre-diabetic subjects. We will assess the surrogate markers of ageing (leukocyte telomere length and telomerase activity) and the expression of longevity genes SIRT1, p66Shc, p53 and mTOR in peripheral blood mononuclear cells (PBMCs) before and after 6 months of metformin treatment.

DETAILED DESCRIPTION:
Research methodology and outcomes measures:

1. Clinical History and Examination: Clinical history and blood pressure.
2. Body mass Index: BMI will be calculated by using formula weight (Kg)/height (m2).
3. Anthropometric Assessment: All circumferences (waist, hip, mid-thigh, mid arm and neck) and skinfolds (biceps, triceps, anterior axillary, subscapular, suprailiac, lateral thoracic and thigh) measurements will be taken. All the measurements will be repeated three times at same position and conditions.
4. Body Composition: Body composition will be measured through multi-frequency bioelectrical impedance (MF-BIA; InBody 770, Cerritos, CA, USA) Visit-2 (Day 90) Visit-3 (Day 180) Compliance check Enrolment of prediabetes subjects (BMI>25kg/m2) (n=112) Investigations: Fasting blood glucose, IGT (2h post-oral glucose load (75g) and HBA1c Group-I: Metformin Group (n=56) Group-II: Placebo Group (n=56) Final Analysis Measurements same as in visit 1 Baseline investigations: Clinical and dietary profiles, blood pressure, anthropometric assessments [body mass index, circumferences (waist, hip, mid-thigh, mid-arm and neck) and skinfolds (biceps, triceps, sub scapular, suprailiac, thigh, lateral thoracic and calf)], body fat, handgrip muscle strength, glycemic and lipid profile other metabolic parameters, fasting serum insulin, C-peptide and HOMA-IR,leukocyte telomerase length and telomerase activity and gene expression of SIRT1, mTOR, p53, p66Shc genes.

   Randomization: Visit 1 (Day 0) Screening Diet and exercise (run in two weeks) 5
5. Handgrip Muscle Strength: Grip strength will be measured using a Jamar Analogue Hand Dynamometer with participants seated, their elbow by their side and flexed to right angles, and a neutral wrist position, the dynamometer handle position II and provision of support underneath the dynamometer.
6. Biochemical measurements: The blood sample shall be drawn after 12 hours overnight fast, subject having taken normal diet in the previous three days. A 75-g OGTT will be performed. Blood samples shall be analyzed for following; blood glucose, A1C, lipids, fasting insulin, C-peptide, Homeostasis Model Assessment (HOMA)- Insulin Resistance (IR), and HOMA- Beta (ß%) and serum glucagon levels.
7. DNA Isolation and Quantification: DNA will be separated from peripheral blood mononuclear cells using the QIAamp DNA extraction kit (Qiagen, Hilden, Germany) and will be stored at -20oC for future experiments. After DNA isolation, the DNA samples will be quantified and diluted to 50 ng/μL. The concentration and quality of DNA will be both measured by using a nanodrop (Nanodrop Technologies, Wilmington, NC, USA) and samples will be included for analysis all will have an optical density ratio A 260/A280> 1.8. h) Measurement of Leukocyte Telomere Length: LTL will be analysed with a quantitative polymerase chain reaction (qPCR) based technique that compares telomere repeat sequence copy number (T) to a reference single copy-gene copy number (S). The telomere length for each sample will be estimated using the telomere to single copy gene ratio (T/S ratio) with the calculation of ΔCt [Ct (telomere)/Ct(single gene)]. T/S ratio for each sample (x) will be normalized to the mean T/S ratio of the reference sample [2-(ΔCtx-ΔCtr) = 2-ΔΔCt], which will be used for the standard curve, both as a reference sample and as a validation sample.

i) Gene expression by real-time PCR: Total RNA will be extracted using aRNeasy Mini Kit, (QIAGEN) cDNA and synthesized with an iScript cDNA synthesis kit (Bio-Rad, USA). Q-PCR assay will be performed in a Thermal Cycler (iCycler iQ5, Bio-Rad, Hercules, CA). Primers for Sirt1, p66Shc, p53, and mTORwill be designed from sequences derived from the GenBank database using Primer 3 (Whitehead Institute, Massachusetts, USA) and Operon's Oligo software (Operon, California, USA), purchased from Eurofins MWG (Ebersberg, Germany). The comparative threshold cycle method (ΔΔCq), which compares differences in the threshold cycle values between groups, will be used to obtain the relative fold change of gene expression.

ELIGIBILITY:
Inclusion Criteria:

Age: 30-60 years Both genders (male and female)

Diagnosis of pre-diabetes, defined as:

Impaired Fasting Glucose (IFG): Fasting plasma glucose 100-125 mg/dL AND/OR Impaired Glucose Tolerance (IGT): 2-hour plasma glucose 140-199 mg/dL after 75 g oral glucose tolerance test (OGTT)

IGT is mandatory (i.e., every participant must have IGT, even if IFG is also present)

Exclusion Criteria:

Type 1 diabetes mellitus Type 2 diabetes mellitus Pregnancy or lactation Hypoglycemia (blood glucose <70 mg/dL) after medication Acute or chronic inflammatory diseases Immunological diseases (e.g., autoimmune diseases) History of organ transplantation Current or recent steroid therapy Uncontrolled arterial hypertension Known allergy or intolerance to metformin Major surgery or cardiovascular events (e.g., myocardial infarction, stroke) within the last 3 months

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Leukocyte telomerase length | 06 months
  Leukocyte Telomere Length Measurement: LTL was analyzed using quantitative polymerase chain reaction (qPCR), comparing telomere repeat sequence copy number (T) to a reference single-copy gene (S). Relative fold changes in gene expression will be determined using the comparative threshold cycle method (ΔΔCq), comparing differences in threshold cycle values between groups.
Telomerase activity | 06 months
  Telomerase activity was done by ELISA method

SECONDARY OUTCOMES:
Expression of longevity genes SIRT1, p66Shc, p53 and mTOR | 6 MONTHS
  Total RNA will be extracted using aRNeasy Mini Kit, (QIAGEN) cDNA and synthesized with an iScript cDNA synthesis kit (Bio-Rad, USA). Q-PCR assay will be performed in a Thermal Cycler (iCycler iQ5, Bio-Rad, Hercules, CA). Primers for Sirt1, p66Shc, p53, and mTORwill be designed from sequences derived from the GenBank database using Primer 3 (Whitehead Institute, Massachusetts, USA) and Operon's Oligo software (Operon, California, USA), purchased from Eurofins MWG (Ebersberg, Germany). The comparative threshold cycle method (ΔΔCq), which compares differences in the threshold cycle values between groups, will be used to obtain the relative fold change of gene expression.

OTHER OUTCOMES:
Weight | 06 month
  Body weight was done by standard weight machine
Height | 06 months
  Height was done by slandered hight scale
Body Mass Index | 6 MONTHS
  BMI by using weight in kilograms (kg) divided by the square of height in meters (m2).
Circumferences | 06 months
  Measurement of circumferences (waist, hip, mid-thigh, mid-arm and neck) was measured with a flexible, non-stretchable tape measure
Skinfold thickness | 06 months
  Skinfolds (biceps, triceps, sub scapular, suprailiac, thigh, lateral thoracic and calf) was measured using skinfold calipers
Body Composition | 6 MONTHS
  Measured via MF-BIA (InBody 770, CA, USA).
Handgrip Muscle Strength | 6 MONTHS
  ssessed using a Jamar Dynamometer with elbows flexed.
Fasting and 75g OGTT | 6 MONTHS
  Blood samples were collected after a 12-hour fast for a 75-g OGTT, analyzing glucose
HAB1C | 06 months
  A1C was done by slandered laboratory
Lipids | 06 months
  Lipids were done by RANDOX kit
Insulin | 06 months
  Serum Insulin done by ELISA kit
C-peptide | 06 months
  C-peptide done by ELISA Kits

CONTACTS AND LOCATIONS:
Locations (1):
- Anoop misra, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No